CLINICAL TRIAL: NCT05885009
Title: Real World Clinical Practice Study to Assess the Feasibility and Impact of Liquid Biopsy-based Genomic Profiling on Treatment Decision Making for Patients With Metastatic Prostate Cancer in Spain (SOLTI-2102)
Brief Title: Feasibility and Impact of Liquid Biopsy Genomic Profiling on Treatment Patients With Metastatic Prostate Cancer in Spain (SOLTI-2102)
Acronym: HOPE-PROSTATE
Status: Recruiting | Type: Observational
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Pfizer (Industry); AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry); Advanced Accelerator Applications (Industry); Astellas Pharma Inc (Industry); Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SOLTI-2102
Record Dates: First submitted 2023-05-03; First posted 2023-06-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Prostate Cancer
Keywords: molecular advisory board; molecular tumor board; genomic data; targeted therapy; patient-centric trials
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection and archival tumor tissue collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Liquid Biopsy — Patients with metastatic prostate cancer in disease progression or not receiving active systemic therapy will undergo a liquid biopsy
Genetic: Archival Tumor DNA sequencing — Patients will be prompted to request an archival tumor sample from metastatic origin (preferably) and to send it to the central laboratory for analysis

SUMMARY:
HOPE Prostate is an observational study that aims at promoting research against metastatic prostate cancer by means of collective research led by patients (patient-centric trial). Patients with metastatic prostate cancer living in Spain will voluntarily register and fulfil their journey in the study through the study's digital tool. Mainly they are prompted to answer questionnaires about their disease, and to provide a blood sample and an archival tumor biopsy. In HOPE Prostate these samples will be genomically analyzed and every patient case will be presented in a multidisciplinary molecular advisory board (MAB). The MAB will issue a plain report explaining the significance of the results and will try to enumerate future therapeutic options that match patient history and his genomic profile. Finally, patients will have to answer short follow-up questionnaires twice a year for 3 years.

The study data will allow us to advance implementing precision medicine to improve the management of current and specially future metastatic prostate cancer patients.

DETAILED DESCRIPTION:
HOPE PROSTATE - SOLTI-2102 is a national, prospective, real-world clinical practice study for patients diagnosed with metastatic prostate cancer (mPC) who are about to receive, or receiving, or completed treatment for advanced disease under standard clinical practice conditions, regardless of where they are receiving their medical care (academics vs community practices).

Patients will lead their own inclusion and, participation, and self-provide follow-up data in the study through a digital tool that will guide them in every step of the journey. The digital tool will collect general patient characteristics and demographics data, informed consent, disease characteristics, diagnostic tools employed along their oncological history, sample collection dates (for tissue,blood and saliva), genetics and tumor mutations, treatment history, patient's expectations and perceptions with regards to the process of undergoing genomic tumor testing and clinical trial experience from patients living with mPC. Moreover, when patients involve their physicians, they will receive notifications from the platform with molecular reports and an invitation to participate in the periodic Molecular Advisory Boards of the study (MAB).

The study will be in accordance with the Declaration of Helsinki and Good Clinical Practice Guidelines and applicable regulatory requirements. Approval of the study protocol will be from an Independent Ethics Committee (IEC).

Patients will request to participate in HOPE-PROSTATE through the study website and a personal session in the digital tool, will be created. Then:

* In a short inclusion questionnaire patients will introduce some demographic and medical data, and if available, medical reports.
* A medical monitor will validate that the inclusion and exclusion criteria are met and will contact patients to explain the study procedures, objectives and answer questions.
* Upon validation, patients will be contacted through the digital tool to give their informed consent or alternatively in paper (at a partner local laboratory).
* After informed consent validation, the digital tool will inform them of the steps to follow to proceed with their patient journey.
* Patients will fill out a short questionnaire to assess their pre-test expectations with regards to anticipated implications of testing and motivations to undergo testing.
* Before results obtention, patients will be required to complete a more extensive questionnaire about their medical history to use it at the Molecular Advisory Board (MAB) meeting.

An information letter will be sent to all patients to be forwarded to their treating physician to be aware of the HOPE-PROSTATE study objectives. Moreover, upon patient's consent, treating physicians will be invited to be registered in a database to be aware of testing progress, receive molecular results and participate in the periodic MAB.

Upon inclusion, patients will be instructed through the digital tool to attend the closest local partner laboratory to perform the necessary blood draw at an appropriate time. In addition, a letter to request the most recent tumor tissue sample at his hospital will be provided; we anticipate collecting tumor tissue samples from at least 80 included patients.

At partner local laboratory:

* Patient may have the possibility to sign the paper study Informed Consent Form if digital signature is not possible.
* Blood samples will be collected (at the time of disease progression).
* Patients will hand over their tumor blocks, previously collected from the local hospitals. At the same time, a saliva sample will be collected.

At the time of documented disease progression and before the initiation of a subsequent line of therapy, patients will be instructed to contact SOLTI to organize their blood sample collection at the closest venue of the partner laboratory. The sample will be sent to the GuardantHealth central laboratory in Redwood City, California. A second blood sample from the same extraction will be shipped to the study central laboratory at Vall d'Hebron Institute of Oncology (VHIO) for complementary analyses.

While we anticipate most mPC patients would join the study in the castration-resistant setting, we plan for a subgroup analysis among patients who join the study at first diagnosis of metastatic, hormone-naïve disease. Patients with metastatic hormone-naïve disease will be included if the blood sample can be collected within 4 weeks from the start of luteinizing hormone releasing hormone antagonist (LHRHa) therapy, although ideally the sample should be collected even before LHRHa initiation. After enrolling 30 hormone-naïve disease patients, we will conduct a feasibility analysis based on the circulating tumor DNA (ctDNA) detection rate (considering an expected detection rate above 80%). If this approach is feasible, the subgroup of patients with metastatic hormone-naïve disease will continue to recruit up to a maximum of 100 patients.

Samples will undergo plasma-based Next Generation Sequencing panel using the "GuardantOMNI" panel test which is a diagnostic system based on the sequencing of 500 genes, as well as the determination of biomarkers that include microsatellite instability (MSI), tumoral mutational burden (TMB) and Homologous Recombination Deficiency (HRD) score. Molecular reports will be generated and sent to the patient physician (if involved), then these data will be discussed at the MAB and a MAB report with molecular data interpretation and a therapeutic recommendation (if there is any) will be send to the patient.

In certain populations of special interest, a repeated ctDNA analysis at a later timepoint will be considered after the MAB evaluation:

* Patients with BRCA gene or HRD pathway alterations who have undergone the test before targeted treatment and develop secondary resistance to PARP inhibitors.
* Patients who have undergone ctDNA prior to exposure to both docetaxel and androgen receptor-targeted agents (ARTA) (SoC Treatments) will be invited to be tested again after progression to these SoC agents to determine the possibility of discovering new therapeutic targets.

At least 80 tumor tissue samples from archival core biopsies or surgical specimens preferably metastatic will undergo genomic characterization. Samples will be sent by participating patients or through treating institutions upon patient's request.

Formaline-fixed paraffin embeeded (FFPE) blocks will be assessed at VHIO by a pathologist and H&E slides will be digitalized. Samples with sufficient tumor content will undergo DNA extraction, quantification and quality control. The obtained DNA will be divided for two downstream applications:

1. All samples will undergo targeted sequencing using a previously validated capture-based panel including >400 genes (mutations, Copy Number Alterations, TMB) at VHIO laboratories and a genomics report will be generated.
2. For those samples with enough DNA quality and quantity after completing the study related targeted sequencing, remaining DNA will be used for retrospective whole exome or whole-genome sequencing (WGS) analysis using modified protocols optimized for FFPE samples for exploratory comparative analysis .

Patients will always have the possibility of getting their treating physician involved in their study participation at any point along the journey which will be recommend by the sponsor. Physicians will be invited to register in a database to inform them most efficiently. They will receive the molecular reports generated and will be invited to participate in the periodic MAB periodic meetings. When the patient case is presented, they will have the opportunity to do so. An informative letter will be provided to all patients so they can share it with their doctors at the time of inclusion.

Besides the study per se, HOPE PROSTATE-SOLTI-2102 educational program for Health Care Professionals (HCP) will focus on physicians treating mPC although their patients participate or not in the investigational part of the study. The two main educational initiatives will be: the Molecular Advisory Board (MAB) meetings and the Initial Educational Meeting.

Upon genomics data availability, patients will have the possibility to update their medical history record through a questionnaire in the platform. Using mPC patient clinical and molecular data a SOLTI dedicated team will prepare the periodic MAB meetings to discuss the cases with new genomics reports available to highlight the potential Scientific relevance of the molecular findings according to patient's clinical progression and discuss potential targeted therapies that could fit each of the cases. The MAB will complement the genomic reports with a text summarizing their interpretation of the results and if possible, the potential future therapeutic strategies that could be considered according to patient profile. We aim at generating a space where mPC HCP can learn about the emerging strategies in mPC management, how to interpret genomics data and embrace a fruitful debate to promote continuous learning about molecular alterations and training on how to use the newly available tools in the clinics. MAB meetings will be scheduled once or twice a month and when possible: they will be complemented with brief educational lectures addressing relevant hot topics in PC management.

Three months after the MAB final report is sent, patients would fill out a second questionnaire to notify if the information received was relevant for subsequent treatment decisions. Moreover, they will be required to fill out the questionnaire to assess the fulfillment of their previous expectations.

This Board will be constituted by a multidisciplinary group of experts in PC clinical management (including medical oncologists, urologists and radiation oncologist), cancer genetics, cancer genomics, bioethics, and pathology. The board aims to be representative of the diversity in our country for managing prostate cancer patients. Besides permanent MAB members, physicians treating HOPE PROSTATE study participants will be invited to participate in the discussions about their patients. Moreover, SOLTI will disseminate the MAB meetings, allowing the free attendance of interested HCP from across the nation. With the aim of promoting participation among nation-wide physicians, these meeting will be held in Spanish and using an online platform.

Irrespective of the MAB outcome, all patients' clinical evolutions will be followed. Patients will be asked to self-report follow-up data every 6 months to determine the status of their disease through the digital tool for at least three years.

To reaffirm the patients-centric approach of HOPE PROSTATE-SOLTI-2102, the study will be complemented by a patient empowerment program that will include informative digital video-capsules and video tutorials about precision medicine and the HOPE Prostate project itself. The content from the digital workshop sessions will be available online and the videos will be public and accessible through the study website to facilitate access to information.

Understanding the patient experience is key to deliver patient-centered care. By looking at various aspects of the patient experience (expectations, concerns, attitudes, and knowledge), we aim at improving healthcare respecting the individual patient's preferences, needs and values.

Before pursuing the genomic test, patients will be invited to complete a series of questionnaires (adapted from previous studies), focused on patients' knowledge about genomic testing and their concerns and expectations around how genomic testing may impact the treatment selection and disease managements9. Three months after MAB report delivery, the same questionnaires will be repeated to evaluate the fulfillment of their previous expectations and the overall experience of the patient participating in the study. After this initial post-recommendation questionnaire, shorter follow up questionnaires will be displayed every six months for three years.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients living in Spain.
2. Age ≥18 years.
3. Signed informed consent before any screening procedure.
4. Metastatic PC of any subtype confirmed both pathologically and radiologically (stage IV disease).
5. The subjects must be about to receive, or receiving, or will have completed treatment for their metastatic disease with any line of treatment in either a clinical trial or the standard of care healthcare setting.
6. Eastern Cooperative Oncology Group (ECOG) 0-1.

Exclusion Criteria:

1. Inability to consent or conform to the processes involved in a clinical study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients diagnosed with metastatic prostate cancer living and being treated in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of a liquid-biopsy based Comprehensive Genomic Panel (CGP) test in the management of mPC patients, following a patient-centric approach | Ongoing basis during 5 years of study duration
  Percentage of patients for whom a liquid biopsy result can be obtained.
To evaluate the impact of a liquid-biopsy based CGP test in the management of mPC patients, following a patient-centric approach | Ongoing basis during 5 years of study duration
  Proportion of patients with a putatively targetable (ESCAT levels I-III) alteration detected.

SECONDARY OUTCOMES:
To describe the genomic landscape of mPC in a real-world population beyond clinical trials using validated targeted sequencing assays in tissue and ctDNA. | Ongoing basis during 5 years of study duration
  Frequency of PC gene mutations in the study population including DNA repair pathways (BRC1/2 inactivating mutations, etc.), genes associated with phosphatidylinositol-3 kinase (PI3K) and cell cycle regulation pathways and others.
To study the feasibility of liquid-biopsy based genomic testing in patient subsets: metastatic hormone-naïve and castration-resistant mPC | Ongoing basis during 5 years of study duration
  ctDNA detection rate in hormone-naïve and castration-resistant mPC.
To study the concordance rate for key genomic alterations between ctDNA and tumor targeted sequencing (in a subset of patients who have both samples available). | Ongoing basis during 5 years of study duration
  * Concordance between ctDNA mutation status and tissue mutation status (specially in Homologous Recombination Repair and other clinically relevant genes).
  * Concordance between ctDNA and tissue TMB calculations.
  * Concordance between ctDNA and tissue Variant Allelle Frequency for given mutations.
To study the clinical impact of genomic testing in terms of matched therapies prescribed from treating physicians. | Ongoing basis during 5 years of study duration
  Percentage of patients who received a matched therapy against an alteration detected by ctDNA and/or tissue targeted sequencing during the follow-up period.
Description Overall Survival (OS) among the included patients | Ongoing basis during 5 years of study duration
  Describe OS from the moment of registration to the death of the patient.
Description Progression Free Survival (PFS) of treatments aimed at identified alterations | Ongoing basis during 5 years of study duration
  Describe PFS with treatments directed to molecular targets identified in ctDNA.

CONTACTS AND LOCATIONS:
Locations (1):
- SOLTI Cancer Research Group, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided